CLINICAL TRIAL: NCT01894958
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose Study of NNZ-2566 in Fragile X Syndrome
Brief Title: A Safety Study of NNZ-2566 in Patients With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neu-2566-FXS-001
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X disorder; Autism
MeSH Terms: conditions — Fragile X Syndrome; Autistic Disorder | interventions — trofinetide; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NNZ-2566 (Experimental): Glycyl-L-2-Methylpropyl-L-Glutamic Acid
  Interventions: Drug: NNZ-2566
- Placebo (strawberry flavored solution) (Placebo Comparator): Strawberry flavored solution and Water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNZ-2566 — Glycyl-L-2-Methylpropyl-L-Glutamic Acid (NNZ-2566) supplied as a lyophilized powder (2g in 50mL vials or 3g in 30mL bottles) for reconstitution with strawberry flavored solution 0.5% v/v in Water for Injection.
  Arms: NNZ-2566
Drug: Placebo — Strawberry flavored solution
  Other Names: Strawberry flavored solution 0.5% v/v in Water for Injection
  Arms: Placebo (strawberry flavored solution)

SUMMARY:
The purpose of this study is to determine whether NNZ-2566 is safe and well tolerated in the treatment of Fragile X Syndrome in adolescent and adult males.

DETAILED DESCRIPTION:
Fragile X Syndrome is a genetically determined neurological disorder in which affected individuals are intellectually handicapped to varying degrees and display a variety of associated psychiatric symptoms. Clinically, Fragile X Syndrome is characterized by intellectual handicap, hyperactivity and attentional problems, autism spectrum symptoms, emotional lability and epilepsy. The epilepsy seen in Fragile X Syndrome is most commonly present in childhood, but then gradually remits towards adulthood. Physical features such as prominent ears and jaw, and hyper-extensibility of joints are frequently present but are not diagnostic. Intellectual handicap is the most common feature defining the phenotype. Treatment for the disorder is symptomatic - focusing on the management of symptoms - and supportive, requiring a multidisciplinary approach.

This study will investigate the safety and tolerability of treatment with oral administration of NNZ-2566 at 35 mg/kg or 70 mg/kg BID in adolescent or adult males with Fragile X Syndrome. The study also will also investigate measures of efficacy during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Fragile X Syndrome with a molecular genetic confirmation of the full FMR1 mutation.

   * Results from previously completed testing are acceptable with written documentation of the genetic results.
   * Results from PCR or Southern blot tests are acceptable
   * Results from cytogenetic testing are not acceptable but subject may be eligible if molecular genetic testing is redone.
   * A full mutation with mosaicism is allowed if:

     * Subject manifests full phenotypic profile of Fragile X syndrome
     * CGG Repeats >200 are detected
     * Southern blot prevails over PCR, if Southern blot shows >200 repeats and PCR results show <200 repeats.
   * The following results would not meet criteria:

     * Deletions
     * Point mutations
     * Mosaicism without detection of >200 CGG repeats or absence of full phenotypic profile in an individual with mosaicism
2. Males, aged 12-45 years
3. Subjects with a Clinical Global Impression - Severity (CGI-S) score of 4 or greater at Screening
4. Subjects with a total score of 30 or greater on the Aberrant Behavior Checklist (ABC) at Screening.
5. Current treatment with no more than 3 psychotropic medications. This includes medications used to treat problems with sleep onset and sleep continuity. Melatonin for difficulties with sleep onset is permissible and is excepted from the count of psychotropic medications. Similarly, anti-epileptic medications are permitted and are not denoted as "psychotropic medications" if they are used for treatment of seizures. Use of anti-epileptics for other indications such as the treatment of mood disorders counts towards the limit of permitted medications. Concurrent use of omega-3 fatty acids is also permissible and does not count towards the allowed number of concomitant psychotropic medications. A complete list of permitted concomitant psychotropic medications can be found in Appendix A.
6. Concomitant medications for chronic medical conditions are permissible. Examples of chronic medical conditions include gastroesophageal reflux disease (GERD) and asthma. Every effort should be made to keep the doses and dosing regimens of these medications stable in the 4 weeks preceding Screening and during the period between Screening and the commencement of study medication.

   1. Permitted psychotropic concomitant medications (except for anti-epileptic medications-see below) must be stable, in terms of dose and dosing regimen, for at least 4 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication.
   2. Anti-epileptic medications must be at a stable dose and dosing regimen for 12 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication
7. Behavioral treatments excluding psychotherapy (see exclusion criteria) must be stable for 4 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication

   a. For each enrollee, every effort should be made to maintain stable regimens of allowed concomitant medications and allowed behavioral therapies from the time of commencement of single-blind study medication until the last study assessment.
8. Sufficient expressive language capabilities to complete the Expressive Language Sampling Task.
9. Individuals with a history of seizures should have a stable pattern of seizure activity in the 3 months preceding Screening.

Exclusion Criteria:

1. Treatment within the two weeks prior to Screening with monoamine (MAO) inhibitors, lithium, minocycline, acamprosate, racemic baclofen, investigational metabotropic glutamate receptor subtype 5 (mGluR5) medications, d-cycloserine, oxytocin, carbetocin, tricyclic antidepressants and bupropion.
2. Patients planning to commence psychotherapy, including cognitive behavior therapy (CBT), during the period of the study or those who had begun psychotherapy, including CBT, within 6 weeks prior to Screening.
3. History of, or current, cardiovascular, renal, hepatic, respiratory and/or gastrointestinal disease, which may interfere with the absorption, distribution, metabolism or excretion of the study medication, or which may interfere with the interpretation of the safety/tolerability or efficacy of the study medication.
4. History of, or current cerebrovascular disease or clinically significant brain trauma.
5. History of, or current clinically significant endocrine disorder, e.g. hypo or hyperthyroidism, or diabetes.
6. History of, or current malignancy.
7. Current major depressive disorder (patients have to be free of the most recent episode for 3 months prior to enrollment).
8. History of a DSM-5-defined substance use disorder in the 3 months prior to Screening.
9. Clinically significant abnormalities in safety laboratory tests, vital signs or ECG, as measured at Screening.
10. QT/QTcF Exclusions (any of the following):

    * QTcF > 450 msec. Three ECGs should be obtained at the time of Screening, 5 minutes apart from each other, and the results should be averaged.
    * History of risk factors for torsade de pointes (e.g. heart failure, clinically significant hypokalemia or hypomagnesemia, or a family of long QT syndrome).
    * A serum potassium at screening <3.0 mmol/L.
    * QT/QTcF prolongation previously or currently controlled with medication, in which normal QT/QTcF intervals could or can only be achieved with medication
    * Current treatment with other medications that have demonstrated QT/QTc prolongation and have this risk described in the Warnings and Precautions section of their Prescribing Information
11. Patients with significant hearing and/or visual impairments that may affect their ability to complete the test procedures.
12. Current treatment with insulin
13. Hgb A1C values outside of the normal reference range at Screening
14. Current or past treatment with insulin like growth factor IGF-1
15. Current or past treatment with growth hormone
16. Enrollment in another clinical trial within the 30 days preceding Screening
17. Previously randomized in this clinical trial
18. Allergy to strawberry

Ages: 12 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | Through to Day 56
  Incidence of adverse events (AE), including Serious adverse events (SAE), will be evaluated between the two NNZ-2566 doses and placebo. Incidence of AEs from randomized dosing through to Day 56 post randomization. Incidence of SAEs from randomization through to Day 56 post randomization.

SECONDARY OUTCOMES:
Physiological changes | Baseline through to Day 56
  Serum levels and changes of standard hematology, and chemistry parameters (including thyroid function) will be calculated from Baseline through to Day 56. Fundoscopy and tonsil size will be documented at Baseline, and Days 14, 28, 42 and 56. Flow cytometry will be used to assess the phosphorylation status of the enzymes Akt and extracellular signal-regulated kinase (ERK) in peripheral lymphocytes, on blood samples obtained on Days 14, 28, 42 and 56. Electrocardiogram (ECG) will be assessed at Screening, Days 14, 21, 28, 35, 42 and 56.
Behavior | Baseline through to Day 56
  Symptom severity according to the Fragile X Symptom Rating Scale, Clinician Domain Specific Top Three Concerns-VAS, Aberrant Behavior Checklist (ABC), Vineland Adaptive Behavior Scale (VABS), Child and Adolescent Symptom Inventory-Anxiety Scale (CASI-16), Children's Yale-Brown Obsessive Compulsive Scale (CYBOCS-PDD), Expressive Language Sampling and Clinical Global Impression of Severity (CGI-S).
Global and Functional outcome Measures | Baseline through to Day 56
  Global outcome as measured by the change in scores in the Clinical Global Impression - Severity and Improvement scales (CGI-S and -I) and the KiTap measure of cognition from baseline, during treatment, and post treatment.
  Global and Functional outcome as measured by changes in scores in the Fragile X Symptom Rating Scale, Clinician Domain Specific Top Three Concerns-VAS, Caregiver Top Three Concerns (related to the subject's Fragile X syndrome) as assessed via a Visual Analogue Scale (VAS), CASI-20, CYBOCS-PDD, Aberrant Behavior Checklist (ABC), Vineland Adaptive Behavior Scales (VABS) and Expressive Language Sampling will be assessed during treatment.

OTHER OUTCOMES:
Pharmacokinetics | During treatment
  The following pharmacokinetic measures will be calculated from NNZ-2566 concentrations in whole blood: Cmax (Peak), Cmin (trough), C0-6 at steady state, and area under the curve (AUC).
Computerized eye-tracking | Baseline through to Day 56
  Computer-based eye tracking assessments will be done on Days 14, 28 and 42.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Berry-Kravis, MD, Principal Investigator — Rush University Medical Center; Joseph Cubells, MD, PhD, Principal Investigator — Emory University; Alexander Kolevzon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Nicole Tartaglia, MD, Principal Investigator — Children's Hospital Colorado; Jean Frazier, MD, Principal Investigator — University of Massachusetts, Worcester; Shivkumar Hatti, MD, Principal Investigator — Suburban Research Associates; Craig Erickson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Thomas Challman, MD, Principal Investigator — Autism & Developmental Medicine Institute Geisinger Health System; Kevin Sanders, MD, Principal Investigator — Vanderbilt University Medical Center; Diane Treadwell-Deering, MD, Principal Investigator — Baylor College of Medicine; Jeffrey Innis, MD, Principal Investigator — University of Michigan; Howard Needleman, MD, Principal Investigator — University of Nebraska; Steve Skinner, MD, Principal Investigator — Greenwood Genetic Center; Bryan King, MD, Principal Investigator — Seattle Children's Hospital; Randi Hagerman, MD, Principal Investigator — UC Davis MIND Institute; Robert Findling, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (17):
- United States (17):
  - UC Davis MIND Institute, Sacramento, California
  - Children's Hospital Colorado, Denver, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Nebraska, Omaha, Nebraska
  - Mount Sinai School of Medicine, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Autism & Developmental Medicine Institute Geisinger Health System, Lewisburg, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Berry-Kravis E, Horrigan JP, Tartaglia N, Hagerman R, Kolevzon A, Erickson CA, Hatti S, Snape M, Yaroshinsky A, Stoms G; FXS-001 Investigators; Glass L, Jones NE. A Double-Blind, Randomized, Placebo-Controlled Clinical Study of Trofinetide in the Treatment of Fragile X Syndrome. Pediatr Neurol. 2020 Sep;110:30-41. doi: 10.1016/j.pediatrneurol.2020.04.019. Epub 2020 May 23. PMID 32660869
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov/
- See also: Fragile X Syndrome — http://ghr.nlm.nih.gov/condition/fragile-x-syndrome
- See also: MECP2 duplication syndrome — http://ghr.nlm.nih.gov/condition/mecp2-duplication-syndrome
- See also: PPM-X syndrome — http://ghr.nlm.nih.gov/condition/ppm-x-syndrome
- See also: Renpenning syndrome — http://ghr.nlm.nih.gov/condition/renpenning-syndrome
- See also: tetrasomy 18p — http://ghr.nlm.nih.gov/condition/tetrasomy-18p
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus/
- See also: Drinking Water — http://www.nlm.nih.gov/medlineplus/drinkingwater.html
- See also: Fragile X Syndrome — http://www.nlm.nih.gov/medlineplus/fragilexsyndrome.html
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks